CLINICAL TRIAL: NCT03387514
Title: Functional Microscale Organotypic Assays to Predict Patient Response to Anti-Angiogenesis Therapies
Acronym: UW17104
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination of funding due to low subject enrollment due to change in standard of care systemic therapy which limited available patients treated with anti-angiogenesis or combined immune and anti-angiogenesis therapy for enrollment.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-1343; P30CA014520 (NIH); A539300 (Other: UW Madison); SMPH/RADIOLOGY/RADIOLOGY* (Other: UW Madison); Protocol Version 4/22/2019 (Other: UW Madison)
Record Dates: First submitted 2017-12-22; First posted 2018-01-02 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Renal Cell Carcinoma
Keywords: Clear Cell; Kidney Cancer; RCC
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a single cohort study without randomization or stratification.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-DCFPyL whole body PET/CT scan (Experimental): 18F-DCFPyL whole body PET/CT scan at three time-points
  Interventions: Drug: PSMA-based 18F-DCFPyL PET tracer for PET/CT exams

INTERVENTIONS:
Drug: PSMA-based 18F-DCFPyL PET tracer for PET/CT exams — 18F-DCFPyL whole body PET/CT scan administered at the following timepoints:
  PET1 - Prior to scheduled nephrectomy
  PET2 - to establish a new baseline PET before systemic therapy
  * PET2A - Post-surgery and prior to start of standard of care systemic therapy
  * PET2B - 12-16 weeks from start of first line systemic therapy (immune-based or anti-angiogenic)
  PET3 - If first line systemic therapy did not include anti-angiogenesis therapy and new systemic therapy does include anti-angiogenesis therapy
  * PET3A - Prior to start of additional anti-angiogenesis therapy
  * PET3B - 12-16 weeks from the start of additional anti-angiogenesis therapy
  PET4 - obtained at clinical progression or 2 years following initial systemic therapy
  Other Names: PSMA PET

SUMMARY:
The primary objective of this research is to evaluate response to systemic therapy, including anti-angiogenesis therapy and/or immune-based therapies via 18F-DCFPyL prostate-specific membrane antigen (PSMA)-based positron emission tomography/computed tomography (PET/CT) in patients with metastatic renal cell carcinoma (RCC) and to compare qualitatively with conventional imaging response criteria - Response Evaluation Criteria In Solid Tumors (RECIST 1.1) and histopathological endpoints including isolation, enumeration and staining of Circulating Tumor Cells (CTC).

DETAILED DESCRIPTION:
Response of systemic therapy, including anti-angiogenesis therapy and/or immune-based therapies will be quantified using PSMA-based PET imaging using a novel agent,18F-DCFPyL, as a non-invasive imaging biomarker of tumor neovasculature to functionally monitor renal cell cancer neovasculature in patients undergoing systemic anti-angiogenesis therapy. PSMA PET will be compared with response to anti-angiogenesis therapy using conventional imaging computed tomography(CT)-based RECIST1.1 criteria as well as histopathological endpoints (tumor vascular density, immunohistochemical staining for PSMA and neovascularization (cluster of differentiation(CD)105, CD31). Whole body PSMA PET/CT scans will be obtained at baseline, following adjuvant anti- angiogenic therapy and when the patient becomes refractory to treatment.

The rationale and time points for obtaining PET scans is planned with respect to the typical natural history of metastatic RCC. This project will obtain information from tumors that are responding to anti-angiogenesis therapy and those resistant to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with locally advanced (>/=cT3) or metastatic clear cell RCC as proven by biopsy.
* Adults, 18 years of age or older.
* Surgical candidates who have clinical indication for nephrectomy and standard-of-care biopsy of metastatic disease followed by possible standard of care systemic anti-angiogenesis based treatment regimen
* Have consented to participate in the University of Wisconsin Carbone Cancer Center Biobank.

Exclusion Criteria:

* Patients who have received prior RCC systemic therapies
* Prior history of prostate cancer
* Prior history of any other malignancy within the last 2 years, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and superficial bladder cancer
* Unable to lie flat during or tolerate PET/CT
* Serum creatinine > 2 times the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-12-08 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Cho, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the University of Wisconsin Carbone Cancer Center from December 2018 to June 2021.
Groups:
- 18F-DCFPyL Whole Body PET/CT Scan: PSMA-based 18F-DCFPyL PET tracer for PET/CT exams administered at the following timepoints:
  PET1 - Prior to scheduled nephrectomy
  PET2 - to establish a new baseline PET before systemic therapy
  * PET2A - Post-surgery and prior to start of standard of care systemic therapy
  * PET2B - 12-16 weeks from start of first line systemic therapy (immune-based or anti-angiogenic)
  PET3 - If first line systemic therapy did not include anti-angiogenesis therapy and new systemic therapy does include anti-angiogenesis therapy
  * PET3A - Prior to start of additional anti-angiogenesis therapy
  * PET3B - 12-16 weeks from the start of additional anti-angiogenesis therapy
  PET4 - obtained at clinical progression or 2 years following initial systemic therapy
Period: Overall Study
Arm/Group | 18F-DCFPyL Whole Body PET/CT Scan
Started | 5
PET 1 | 5
Tissue Samples | 4
PET 2A | 0 (Due to change in standard of care system therapy to immune therapy during the course of this trial, patients did not proceed to anti-angiogenesis therapy or combined anti-angiogenesis therapy with immune therapy to allow for PET imaging 2A or further PET imaging timepoints during the follow-up period of this trial.)
PET 2B | 0 (Due to change in standard of care system therapy to immune therapy during the course of this trial, patients did not proceed to anti-angiogenesis therapy or combined anti-angiogenesis therapy with immune therapy to allow for PET imaging 2A or further PET imaging timepoints during the follow-up period of this trial.)
PET 3A | 0 (Due to change in standard of care system therapy to immune therapy during the course of this trial, patients did not proceed to anti-angiogenesis therapy or combined anti-angiogenesis therapy with immune therapy to allow for PET imaging 2A or further PET imaging timepoints during the follow-up period of this trial.)
PET 3B | 0 (Due to change in standard of care system therapy to immune therapy during the course of this trial, patients did not proceed to anti-angiogenesis therapy or combined anti-angiogenesis therapy with immune therapy to allow for PET imaging 2A or further PET imaging timepoints during the follow-up period of this trial.)
PET 4 | 0 (Due to change in standard of care system therapy to immune therapy during the course of this trial, patients did not proceed to anti-angiogenesis therapy or combined anti-angiogenesis therapy with immune therapy to allow for PET imaging 2A or further PET imaging timepoints during the follow-up period of this trial.)
Completed | 0 (Due to change in standard of care system therapy to immune therapy during the course of this trial, patients did not proceed to anti-angiogenesis therapy or combined anti-angiogenesis therapy with immune therapy to allow for PET imaging 2A or further PET imaging timepoints during the follow-up period of this trial.)
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | 18F-DCFPyL Whole Body PET/CT Scan
Number analyzed (Participants) | 5
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 1
  40-49 years | 0
  50-59 years | 1
  60-69 years | 2
  70-79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
PET maximum SUV (SUVmax) [Mean (Standard Deviation); unit: SUV] — PET standardized uptake value (SUV) is defined as:
  SUV = C(T) / (injection dose [MBq]/patient's weight [kg])
  which represents the tumor or tissue radiotracer concentration at a point in time C(T) relative to the total concentration of radiotracer activity in the entire patient (total injected dose of radioactivity per kilogram of the patient's body weight), with body weight used as a surrogate for a distribution volume of radiotracer.
  Maximum SUV (SUVmax) is the maximum or highest radiotracer activity within a defined ROI.
  SUV | 6.60 (3.16)

OUTCOME MEASURES:

1. Primary Outcome: Baseline Tumor FDG PET SUV Data by Disease Type at Baseline
Description: Tumor FDG PET SUV data is provided from baseline PET tumor data. Participants with baseline 18F-DCFPyL PSMA PET/CT prior to surgical nephrectomy and metastatic disease sampling were analyzed based single timepoints for PET SUVmax values of tumor uptake (primary and metastatic disease)
Time Frame: Baseline
Population: Five patients with baseline 18F-DCFPyL PSMA PET/CT prior to surgical nephrectomy and metastatic disease sampling were analyzed based on limited sample size and single timepoints for PET SUVmax values of tumor uptake (primary and metastatic disease).
Measure: Mean (Standard Deviation); unit: SUV
Groups:
- 18F-DCFPyL PET/CT Scan - Primary: Primary Renal Tumor
- 18F-DCFPyL PET/CT Scan - Metastases: Metastatic Lesions
- 18F-DCFPyL PET/CT Scan - Bone Metastases: Bone Metastases
- 18F-DCFPyL PET/CT Scan - Soft Tissue Metastases: Soft tissue metastases
Arm/Group | 18F-DCFPyL PET/CT Scan - Primary | 18F-DCFPyL PET/CT Scan - Metastases | 18F-DCFPyL PET/CT Scan - Bone Metastases | 18F-DCFPyL PET/CT Scan - Soft Tissue Metastases
Number analyzed (Participants) | 5 | 5 | 5 | 5
SUV | 8.78 (3.35) | 5.51 (2.56) | 7.57 (3.43) | 4.63 (1.70)

2. Primary Outcome: Histopathological Endpoints: Immunohistochemical Staining for PSMA
Description: Compare PSMA imaging to histopathological endpoints which include tumor vascular density, immunohistochemical staining for PSMA and neovascularization (CD105, CD31 markers)
Time Frame: Up to 24 months
Population: Data were not collected for Immunohistochemical PSMA staining due to termination of funding for this study due to low accrual (see section on limitation and caveats).
Groups:
- 18F-DCFPyL Whole Body PET/CT Scan: PSMA-based 18F-DCFPyL PET tracer for PET/CT
Arm/Group | 18F-DCFPyL Whole Body PET/CT Scan
Number analyzed (Participants) | 0

3. Primary Outcome: Histopathological Endpoints: Tumor Vascular Density
Description: as for outcome 2
Time Frame: Up to 24 months
Population: Data were not collected for Tumor vascular density due to termination of funding for this study due to low accrual (see section on limitation and caveats).
Arm/Group | 18F-DCFPyL Whole Body PET/CT Scan
Number analyzed (Participants) | 0

4. Primary Outcome: Histopathological Endpoints: Neovascularization Measured by CD105 and CD31 Markers
Description: as for outcome 2
Time Frame: Up to 24 months
Population: Data were not collected for CD105 and CD31 neovascularization due to termination of funding for this study due to low accrual (see section on limitation and caveats).
Arm/Group | 18F-DCFPyL Whole Body PET/CT Scan
Number analyzed (Participants) | 0

5. Secondary Outcome: Measure Therapy Response of Patient Specific uVESSEL (a Micro Scale Organotypic Co-culture Model): Vessel Sprouting
Description: Patient-derived uVESSEL models (from primary & metastatic sites) and incorporating patient-derived immune cells, will be tested for response to anti-angiogenic therapies including pazopanib, sunitinib, cabozantinib, and axitinib. Response will be quantified via multiple endpoints, e.g. vessel sprouting, PSMA expression, cell death.
Time Frame: Up to 24 months
Population: Patient tumor specimen were processed and positively selected for CD31 cells, for endothelial and epithelial cell fractions. Microphysiological models were established using the two cell populations using a mold casting strategy. Models were treated with therapeutic agents after 24 hr in culture and incubated with the agent for 72hr. Imaging with confocal microscopy was used to determine individual sprout numbers. Values were acquired from at least 2 independent experiments.
Measure: Mean (Standard Error); unit: Sprout number
Groups:
- Vessel Sprout Number: Patient 1; Vessel Sprout Number: Patient 2: Number of individual sprout numbers from in-vitro model
Arm/Group | Vessel Sprout Number: Patient 1 | Vessel Sprout Number: Patient 2
Number analyzed (Participants) | 1 | 1
Sprout number
  Vehicle Control | 4.333 (1.211) | 5.364 (0.927)
  Sunitinib | 2.000 (1.155) | 13.330 (2.369)
  Pazopanib | 2.400 (1.140) | 15.330 (3.964)
  Cabozantinib | 3.333 (0.333) | 21.300 (3.512)
  Axitinib | NA (NA) — Not tested | NA (NA) — Not Tested

6. Secondary Outcome: Evaluate the Predictive Power and Validate the uVESSEL Model
Description: Using the clinical, pathological and imaging endpoints, predictive models will e developed using responses to uVESSEL model above. More specifically the objective response (dichotomous endpoint of yes or no) measured using PSMA-based PET/CT will be used as a dependent variable in a logistic regression model with response to uVESSEL model from above as an independent predictor to segregate uVESSEL responses into two groups corresponding to responders and non-responders to anti-angiogenic therapies.
Time Frame: Up to 24 months
Population: Data were not collected to evaluate the predictive power and validation of the uVESSEL model due to termination of funding for this study due to low accrual (see section on limitation and caveats).
Groups:
- uVESSEL Model Predictive Model: PSMA-based 18F-DCFPyL PET baseline imaging cohort
Arm/Group | uVESSEL Model Predictive Model
Number analyzed (Participants) | 0

7. Secondary Outcome: Measure Therapy Response of Patient Specific uVESSEL (a Micro Scale Organotypic Co-culture Model): PMSA Expression
Description: as for outcome 5
Time Frame: Up to 24 months
Population: Data were not collected due to termination of funding for this study due to low accrual (see section on limitation and caveats).
Arm/Group | uVESSEL Model Predictive Model
Number analyzed (Participants) | 0

8. Secondary Outcome: Measure Therapy Response of Patient Specific uVESSEL (a Micro Scale Organotypic Co-culture Model): Cell Death
Description: Patient-derived uVESSEL models (from primary & metastatic sites) and incorporating patient-derived immune cells, will be tested for response to anti-angiogenic therapies including pazopanib, sunitinib, cabozantinib, and axitinib. Response will be quantified via multiple endpoints, e.g. vessel sprouting, PSMA expression, cell death. Two subjects had data collected and were assessed.
Time Frame: Up to 24 months
Population: A version of the models without endothelial cells was generated to evaluate tumor (only) response to therapeutics. To this end, a luminescent reagent was used to assess the amount of ATP in the models, which can be correlated to the number of live cells in the model. Measurements were taken at day 0 and at day 4 (after 72h of treatment) and normalized to account for patient-specific ATP variations. Values were acquired from at least 2 independent experiments.
Measure: Mean (Standard Error); unit: Sprout number
Groups:
- Tumor Response to Therapeutics: Patient 1; Tumor Response to Therapeutics: Patient 2: Tumor only response to anti-angiogenesis inhibitors (ATP cell assay)
Arm/Group | Tumor Response to Therapeutics: Patient 1 | Tumor Response to Therapeutics: Patient 2
Number analyzed (Participants) | 1 | 1
Sprout number
  Vehicle Control | 148.8 (6.838) | 70.67 (3.23)
  Sunitinib | 28.98 (4.86) | 38.38 (2.06)
  Pazopanib | 94.74 (1.62) | 89.46 (2.57)
  Cabozantinib | 54.05 (1.23) | 110.40 (7.05)

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | 18F-DCFPyL Whole Body PET/CT Scan
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Due to change in standard of care system therapy to immune therapy during the course of this trial, patients did not proceed to anti-angiogenesis therapy or combined anti-angiogenesis therapy with immune therapy to allow for further PET or CT maging timepoints during the follow-up period of this trial. Therefore RECIST 1.1 response could not be assessed but PET SUVmax data is provided. Due to low enrollment for this issue, the study funding did not continue to allow for further study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT03387514/Prot_SAP_000.pdf